CLINICAL TRIAL: NCT05048381
Title: miRNA in Sweat, a Novel Digital Biomarker for Detection of Active Tuberculosis
Brief Title: miRNA in Sweat, a Novel Digital Biomarker for Detection of Active Tuberculosis (TB)
Status: Withdrawn | Type: Observational
Why Stopped: Technical challenges during lab sweat analysis lead to run out of funding
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Fachhochschule Nordwestschweiz (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01810; am21Eckstein2
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Active Tuberculosis
Keywords: miRNA; Mycobacterium Tuberculosis; Next Generation Sequencing
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing — Next Generation Sequencing of sweat and whole blood samples for non-coding miRNAs to define biomarkers that enable to differentiate between patients with active tuberculosis, a differential diagnostic disease and healthy individuals.

SUMMARY:
The detection of miRNA (non-coding ribonucleic acid) in the blood in the context of active tuberculosis is an innovative approach to the detection of new disease-specific biomarkers.

The primary goal of this analysis is to define, for the first time, an miRNA fingerprint for tuberculosis in sweat. Samples that were collected as part of the Sweatb Study (NCT03667742) project are examined for the occurrence of disease-specific, non-coding miRNAs to define new biomarkers in the sweat. These biomarkers can be detected non-invasively and will help in the detection of patients with active tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Ability to understand the purpose of the study, provide signed and dated informed consent by patient or his/her legal representative
* In-patients with acute tuberculosis, suspected tuberculosis or other pulmonary diseases (pneumonia, Bronchitis, COPD)

Inclusion criteria Healthy Donors:

* negative for Quantiferon- TB Gold Plus Test or ELISpot

Exclusion Criteria:

* Written rejection of the consent for the further use of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants in the Sweatb study (NCT03667742)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Detection of miRNA (non-coding ribonucleic acid) in sweat | Sweat samples taken at baseline
  Analysis of sweat protein markers in patients with active tuberculosis
Detection of miRNA (non-coding ribonucleic acid) in blood | Blood samples taken at baseline
  Analysis of blood protein markers in patients with active tuberculosis

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, Prof. Dr. med., Principal Investigator — Chief Medical Information Office (CMIO), University Hospital Basel